CLINICAL TRIAL: NCT00389883
Title: Anaesthesia for Supratentorial Tumor Resection : a Double-blind Comparison of Target Plasma Concentration of Propofol-remifentanil and Sevoflurane-sufentanil
Brief Title: Anaesthesia for Supratentorial Tumor Resection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P050320
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Supratentorial Neoplasms
Keywords: supratentorial brain tumors; propofol; sevoflurane; remifentanil; sufentanil.
MeSH Terms: conditions — Supratentorial Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): propofol et remifentanil
  Interventions: Drug: Comparison of two anesthetics protocol
- 2 (Experimental): sevoflurane et sufentanil
  Interventions: Drug: Comparison of two anesthetics protocol

INTERVENTIONS:
Drug: Comparison of two anesthetics protocol — Comparison of two anesthetics protocol

SUMMARY:
This is a double center, multidisciplinary, prospective, randomized, double-blind, with a superiority hypothesis, trial including 100 patients scheduled for resection of a supratentorial brain tumour under general anesthesia.

DETAILED DESCRIPTION:
On the morning of surgery, patients will be randomly allocated to one of the two following groups : target concentration-delivered propofol-remifentanil versus sufentanil-sevoflurane. The primary judgement criterion will be the rapidity of awakening, defined as the time between the cessation of administration of the last anesthetic until extubation. Several secondary judgement criteria related to quality of postoperative recovery and complications will be collected. The hypothesis tested is a 30% reduction of the time necessary to extubate patients after cessation of anesthetic delivery in the propofol-remifentanil group. Based on previous works, using an risk of 20 % and an of 5 %, 100 patients must be included in this study (50 or each group). Statistical analysis will be performed by WILCOXON MANN, WHITNEY and X2 tests based on the type of variables.

The results of this study should provide a first choice anaesthetic regimen to optimize postoperative recovery of neurosurgical patients undergoing resection of supratentorial brain tumours. They will contribute to the improvement in the management of patients suffering from cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for supratentorial brain tumors remove.
* Age : 18 to 75.
* ASA 1 or 2.

Exclusion Criteria:

* Disagree of patient to participate
* Intubation required in the postoperative care unit
* Contraindication of one of the anesthetics used in the study
* Pregnancy
* Craniotomy in the frontal area (no depth of anesthesia monitoring)
* Patient's inability to quantified its pain.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Time from discontinuing anesthesia and extubation. | during 24 hours

SECONDARY OUTCOMES:
Speed of emergence from anesthesia : time from discontinuing anesthesia to spontaneous breathing, opening the eyes, response to simple order and discharge from postoperative care unit. | during 24 hours
Quality of emergence from anesthesia : agitation, postoperative pain, nausea and vomiting, cognitive functions. | during 24 hours
Quality of surgical procedure : Coma glasgow scale, surgical procedure difficulties. | during 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Souhayl DAHMANI, MD,PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (2):
- France (2):
  - Centre Hospitalier Universitaire., Besançon
  - Hopital BEAUJON ASSISTANCE PUBLIQUE, Clichy

REFERENCES:
- [Result] Todd MM, Warner DS, Sokoll MD, Maktabi MA, Hindman BJ, Scamman FL, Kirschner J. A prospective, comparative trial of three anesthetics for elective supratentorial craniotomy. Propofol/fentanyl, isoflurane/nitrous oxide, and fentanyl/nitrous oxide. Anesthesiology. 1993 Jun;78(6):1005-20. doi: 10.1097/00000542-199306000-00002. PMID 8512094
- [Derived] Necib S, Tubach F, Peuch C, LeBihan E, Samain E, Mantz J, Dahmani S; PROMIFLUNIL trial group. Recovery from anesthesia after craniotomy for supratentorial tumors: comparison of propofol-remifentanil and sevoflurane-sufentanil (the PROMIFLUNIL trial). J Neurosurg Anesthesiol. 2014 Jan;26(1):37-44. doi: 10.1097/ANA.0b013e31829cc2d6. PMID 23774117